CLINICAL TRIAL: NCT04859062
Title: The Effect of Applying Xylocaine Gel 2% to the Eye Preoperatively in Pediatrics Undergoing Squint Surgeries on Oculocardiac Reflex Intraoperatively and Postoperative Pain and Agitation: Cohort Study
Brief Title: Lidocaine Gel 2% and Muscle Traction Pain During Squint Surgery in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Principal Investigator, Abeer Samir Salem, Researcher, Research Institute of Ophthalmology, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23334
Record Dates: First submitted 2021-04-08; First posted 2021-04-26 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Squint
Keywords: squint; muscle traction; pain
MeSH Terms: conditions — Strabismus; Pain | interventions — Anesthesia; Control Groups

STUDY DESIGN:
Intervention Model Description: 2 group control and xylocaine gel 2% group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): no lidocaine gel 2% is applied
  Interventions: Other: control group
- lidocaine group (Experimental): the lidocaine gel 2% is applied to the operative eye preoperatively
  Interventions: Drug: lidocaine gel 2%

INTERVENTIONS:
Drug: lidocaine gel 2% — assessing its efficacy in decreasing muscle traction pain,In the operation room, we started inhalational induction of anesthesia with sevoflurane till the patient is deeply anesthetized. In the experimental group, we applied lidocaine gel 2% abundantly below both eyelids of the surgical eye for at least 3 minutes before the surgical incision, while nothing was applied to patients in the control group.
  Other Names: xylocaine gel, topical anesthesia
  Arms: lidocaine group
Other: control group — In the operation room, we started inhalational induction of anesthesia with sevoflurane till the patient is deeply anesthetized. In control group, we didn't apply lidocaine gel 2% to the operative eye .
  Arms: control

SUMMARY:
Assessing the efficacy of lidocaine gel 2% application 10 minutes before surgery on post operative pain and the use of analgesics postoperatively

DETAILED DESCRIPTION:
After inhalational induction of anesthesia and applying the pulse oximeter to the patient's finger but and before cannulating or managing the patient's airway lidocaine gel 2% is efficiently applied to the surgical eye (to give more time for the gel to act without delaying the surgery) then cannulation and laryngeal mask inserted to maintain ventilation properly.

Applying lidocaine gel 2% should be filling the upper and lower 10 minute fornices before disinfecting the eye and starting the surgery

The primary outcome is assessing postoperative pain and need for postoperative systemic analgesia The secondary outcome is to monitor the oculocardiac reflex intraoperatively and the need for intraoperative atropine.

ELIGIBILITY:
Inclusion Criteria:

* age 3 to 12 years
* squint surgery

Exclusion Criteria:

* below 2 years or more than 13

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after recovery in PACU using FLACC score (Face, Leg, Activity, Cry, Condolence) | during surgery
  FLACC (Face, legs, activity, cry, condolence): each parameter will take a score from 0 to 2 and the total of the 5 parameters is a score of pain ; 0 is for no pain and 10 is maximal pain

SECONDARY OUTCOMES:
oculocardiac reflex occurrence during muscle traction intraoperative | during surgery
  bradycardia at muscle traction during surgery

CONTACTS AND LOCATIONS:
Overall Officials: abeer salem, MD, Principal Investigator — research institute of ophthalmology
Locations (1):
- Research Institute of Ophthamology, Giza, Egypt